CLINICAL TRIAL: NCT04617496
Title: An RCT of a Telemedicine Intervention for Hypokinetic Dysarthria in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E3378-R
Record Dates: First submitted 2020-10-29; First posted 2020-11-05 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Dysarthria; Speech therapy
MeSH Terms: conditions — Parkinson Disease; Dysarthria; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined speech and exercise intervention (Experimental): Home-based exercise intervention with interactive automated speech response features that encourage a higher level of speech performance.
  Interventions: Behavioral: Combined speech and exercise intervention
- Control group (Active Comparator): Health education
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Combined speech and exercise intervention — Home-based exercise intervention with interactive automated speech response features
  Arms: Combined speech and exercise intervention
Behavioral: Health education — Provision of general information about a variety of topics
  Arms: Control group

SUMMARY:
Nearly 90% of people with Parkinson's disease have speech and voice disorders that negatively impact their ability to communicate effectively in daily life. This study will test the hypothesis that a combined speech and exercise intervention will improve speech intelligibility in people with Parkinson's disease and speech impairment. This approach would offer an affordable way to continue to both instruct and encourage training by Veterans virtually indefinitely through the remote access technology. These findings may help VA clinicians provide optimal care for the many Veterans with Parkinson's disease and speech impairment.

DETAILED DESCRIPTION:
Background/Rationale The great majority of individuals with Parkinson's disease (PD) develop speech impairments, most of which are grouped together and called hypokinetic dysarthria. Hypokinetic dysarthria is typically characterized by altered prosody (e.g., reduced loudness and pitch variation), phonation (e.g., breathy or harsh voice), and articulation (e.g., imprecise consonants, centralized vowels). Changes in speech may appear early in PD and progress in severity over time. Further, such changes in speech lead to significant declines in functional communication and quality of life. Pharmacological and surgical interventions that alleviate motor symptoms in PD are largely ineffective or sometimes even detrimental for speech.

Objectives Based on results from a preliminary study, the investigators propose to conduct a pilot randomized, controlled trial in patients with hypokinetic dysarthria in PD to assess the potential effectiveness of a novel home-based exercise intervention with interactive automated speech response features that encourage a higher level of speech performance. The investigators hypothesize that patients in the intervention program will improve in speech intelligibility and self-perceived communication ability over 6 months, as compared with patients in a health education program.

Methods A total of 104 community-dwelling Veterans with hypokinetic dysarthria in mild-to-moderate PD will be randomly assigned to the exercise intervention or to the health education control. The investigators will test the effects of the intervention at 6 months for the outcomes speech intelligibility and self-perceived communication ability.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of idiopathic Parkinson's disease (PD)
* At least 2 of the 3 cardinal signs of PD (resting tremor, rigidity, bradykinesia)
* Response to dopaminergic medication
* Hypokinetic dysarthria

Exclusion Criteria:

* Angina pectoris
* History of myocardial infarction (MI) within 6 months
* History of ventricular dysrhythmia requiring current therapy

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combined Speech and Exercise Intervention | Control Group
Started | 50 | 54
Completed | 45 | 50
Not Completed | 5 | 4
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Speech and Exercise Intervention | Control Group | Total
Number analyzed (Participants) | 50 | 54 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (5.5) | 73.5 (6.5) | 74.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 54 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White, Non-Hispanic | 50 | 53 | 103
  Race/Ethnicity: Black | 0 | 1 | 1
Speech Intelligibility [Mean (Standard Deviation); unit: units on a scale] — Speech intelligibility is the degree to which spoken language can be understood by a listener and measured by the percentage of words understood from a recording of a participant reading a random set of 11 sentences from the Assessment of Intelligibility in Dysarthric Speech Sentence Intelligibility Test stimulus bank. Possible scores range from 0 (no words understood) to 100 (all words understood). (please see outcomes section for full description)
  units on a scale | 48.7 (23.0) | 46.5 (18.4) | 47.7 (20.8)
Communication Effectiveness Score [Mean (Standard Deviation); unit: units on a scale] — Possible scores range from 10 (worst rated effectiveness) to 100 (best rated effectiveness).
  units on a scale | 50.6 (18.2) | 57.5 (14.1) | 54.2 (16.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Speech Intelligibility at 6 Months
Description: Speech intelligibility is the degree to which spoken language can be understood by a listener. It is measured by the percentage of words that are understood from a recording of a participant reading a random set of 11 sentences from the Assessment of Intelligibility in Dysarthric Speech Sentence Intelligibility Test stimulus bank. Native speakers of American English listened to these recordings to assess speech intelligibility. These listeners were between the ages of 18 and 35 with no history of speech, language, or hearing disorders or experience rating speech. Each listener was provided with one sentence from each study participant's recording. Listeners were asked to transcribe each sentence to the best of their ability. Their transcriptions were compared with the actual sentences to calculate the percentage of words that were understood. Possible scores range from 0 (no words understood) to 100 (all words understood). Change = (6-month score - Baseline score)
Time Frame: Baseline and 6-month Follow-up
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Combined Speech and Exercise Intervention | Control Group
Number analyzed (Participants) | 40 | 37
score on a scale | 0.25 [-23.5 to 28.6] | -4.78 [-45.9 to 24.4]
Statistical Analysis 1: Comparison: Combined Speech and Exercise Intervention vs Control Group; Test type: Superiority; p = 0.13, Mixed Models Analysis; Mean Difference (Net) = 5.0, Standard Error of Mean 3.3

2. Secondary Outcome: Change in in Self-perceived Communication Ability Measured Via the Communication Effectiveness Index (CETI-M) at 6 Months
Description: CETI-M is a self-reported instrument assessing participants' communicative effectiveness in 10 different speaking situations (e.g., in noisy environments; over the phone) on a 10-point Likert scale, where 1 = not effective and 10 = extremely effective. Possible scores range from 10 (worst rated effectiveness) to 100 (best rated effectiveness).
  Change = (6-month score - Baseline score)
Time Frame: Baseline and 6-month Follow-up
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Combined Speech and Exercise Intervention | Control Group
Number analyzed (Participants) | 45 | 50
score on a scale | 6.8 [-33.1 to 57.0] | -6.4 [-55.0 to 32.0]
Statistical Analysis 1: Comparison: Combined Speech and Exercise Intervention vs Control Group; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Combined Speech and Exercise Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 2/50 | 1/54
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/54
Other Adverse Events (participants affected / at risk) | 0/50 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT04617496/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT04617496/ICF_000.pdf